CLINICAL TRIAL: NCT04815980
Title: Impact of Pilates Mat-Based Exercises on Knee Kinematics During Running
Brief Title: Impact of Pilates on Running Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, Alexis Ortiz, Professor, University of the Incarnate Word
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A4160108
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Strength; Exercise; Knee Injuries
Keywords: Pilates; Running; Knee
MeSH Terms: conditions — Motor Activity; Knee Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups randomized; no-exercise control vs. Pilates exercise group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group performed no Pilates intervention. They continued with their typical activities of daily living.
- Pilates (Experimental): Participants in this group performed a 30 minute mat-based Pilates intervention 3 times/week for 12 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Home-based mat-based Pilates intervention 3 times a week for 12 weeks prepared by a certified Pilates instructor.
  Arms: Pilates

SUMMARY:
INTRODUCTION: Core strengthening, balance, and flexibility programs such as Pilates have been advocated to affect running mechanics and prevent lower extremity injuries positively. The purpose of this study was to assess the effects of a 12-week mat-based Pilates exercise program on dynamic knee valgus alignment in runners.

METHODS: Thirty-four young male and female adults performed a running protocol at baseline. The protocol consisted of the participants running on a treadmill at a constant five miles per hour (mph) for four minutes. Post-examination, participants were randomly assigned to a Pilates or control group (n=16 and n=18, respectively). A certified Pilates instructor gave the Pilates group a 12-week home-based program. To ensure participants in the Pilates group performed exercises correctly, the Pilates instructor conducted the first session, and provided feedback to each participant. Participants in both groups performed the same running testing protocol every four weeks. Knee valgus was measured as the medial displacement of the knee joint center during the running stance phase. Repeated measures Analysis of Variance (RepANOVA) was calculated at baseline and 4-, 8-, and 12-weeks post examinations to compare knee valgus during running.

DETAILED DESCRIPTION:
Study Design and Participants A 12-week randomized controlled trial using a mat-based Pilates core-strengthening exercise program was conducted involving thirty-four young, healthy adults. Twenty men (mean ± SD; height: 171.77 ± 9.42 cm; weight: 72.59 ± 8.99 kg; BMI: 24.99 ± 2.10 kg/m2) and fourteen women (mean ± SD; height: 158.46 ± 2.96 cm; weight: 53.70 ± 2.45 kg; BMI: 21.81 ± 1.37 kg/m2) completed this study. All participants were over 18 and signed a written informed consent document approved by the Institutional Review Board. Inclusion criteria included no history of injury in the preceding six months, no history of lower extremity surgeries, and a generally healthy state. Before involvement in the main trials, each participant's height, body mass, leg length, pelvis, knee, and ankle width were measured according to the motion analysis software computerized model (Vicon Plugin Gait Model, Vicon Motion Inc., Denver, CO).

Procedures Participants reported to the laboratory having refrained from strenuous exercise during the preceding 48 hours. A running protocol was conducted four times during this study: at baseline, and at the fourth, eighth, and twelfth weeks. Participants underwent a standardized warm-up session running at four miles per hour (mph) on a treadmill for five minutes before progressively increasing the intensity to five mph without any inclination for another four minutes. To measure dynamic knee valgus during each session, a 3-dimensional high-speed (240 Hz) system (Vicon Motion Inc., Denver, CO) was used during the running protocol, emphasizing the running cycle's stance phase to measure medial knee displacement. For each participant, 3D kinematics were recorded for the dominant leg throughout the stance phase during the running protocol execution. The dominant leg was defined as the preferred leg to perform a single leg jump. Medial knee displacement was defined as the medial trajectory difference traveled by the knee joint center from initial contact to push-off, identified by two footswitches (500Hz; Delsys, Inc, Boston, MA) placed on the plantar aspect of the calcaneus and hallux. Three-dimensional data and pressure from the footswitches were real-timed synchronized in the motion analysis software (Vicon Nexus software, Vicon Motion Inc., Denver, CO).

Once baseline measurements were recorded, the participants were randomly assigned to either a home-based Pilates intervention or a control group. The Pilates intervention consisted of a warm-up, seven strengthening exercises, and a cool-down. The frequency of the program was three times a week, performing each exercise once for 15 repetitions. Participants in the Pilates group performed their first session with a certified Pilates instructor to ensure appropriate technique was performed. The control group was encouraged to continue their daily routine and not engage in additional physical activity or exercise. At the fourth and eighth weeks, the Pilates program's difficulty level increased by progressing to more challenging exercises.

Data Analysis T-tests were performed at baseline for anthropometrics and valgus variables to ensure both groups were homogenous. A 2 x 4 (group x time) repeated measures ANOVA (RepANOVA) was used to evaluate dynamic knee valgus changes. Group by time interaction and within and between main effects were separately assessed regardless of the interaction being significant based on recommendations by Wei et al. 2012 (Wei et al., 2012). Given the pilot nature of this investigation, an alpha level of p ≥ 0.05 was considered statistically significant for all analyses. SPSS version 26 (IBM SPSS, Armonk, New York) was used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* generally healthy state

Exclusion Criteria:

* no history of injury in the preceding six months
* no history of lower extremity surgeries

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2010-09-10 (Actual); Study Completion 2010-09-10 (Actual)

PRIMARY OUTCOMES:
Knee Valgus | 12 weeks
  Medial displacement of the knee from the moment of foot strike to push-off

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ortiz, PhD, Principal Investigator — University of the Incarnate Word
Locations (1):
- University of The Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No